CLINICAL TRIAL: NCT00094874
Title: A Double-Blind, Randomized Study of Puncturing Versus Non-Puncturing Acupuncture for the Treatment of Interstitial Cystitis Symptoms
Brief Title: Acupuncture for the Treatment of Interstitial Cystitis (IC) Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Mary Elizabeth Groff Surgical Medical Research and Education Charitable Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 801685
Record Dates: First submitted 2004-10-27; First posted 2004-10-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Interstitial Cystitis
Keywords: pelvic pain, bladder pain, urgency, frequency, nocturia
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain; Nocturia | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Acupuncture is a form of Chinese medicine that has been in existence for more than a thousand years. This clinical trial performs two types of acupuncture on traditional 'bladder' points to determine if one type demonstrates improvement over the other. In the first type needles stimulate acupuncture points on the skin, and in the second type the needles penetrate through the skin similar to how acupuncture is usually performed. The technique is done through shields so that people will not know what type of acupuncture they receive.

Patients must have at least moderately severe disease as determined by a urologist. They must be willing not to change their medical regimen for the duration of the trial. Patients will receive twelve treatments over six to twelve weeks. They will be asked to fill out symptom questionnaires and bladder diaries at regular intervals to monitor change. All treatment is free of charge, and patients who complete the trial will receive a small stipend.

DETAILED DESCRIPTION:
Patients eligible for enrollment include:

* Age 18-65 years
* Symptomatic IC for at least six months
* Urinary frequency of at least eleven voids in a 24 hour period
* A self-rated global discomfort score of 4 or greater on a 0-10 scale

Patients may not be enrolled who have a history of chronic bladder disease or pelvic disease including cancer, calculi, infection or complications of nervous system disease or diabetes. They must be on no blood thinning agents or have had any recent medication changes or bladder procedures.

After screening physical examination and history-taking, patients will be asked to fill out standard symptom questionnaires. They will be given a bladder diary to fill out for the 24 hours prior to their first acupuncture treatment which will be scheduled within a week.

Patients will be asked to return from once- to twice-weekly for a total of twelve treatments. Patients will complete a bladder diary before each treatment and a questionnaire form before every other visit. The same questionnaire will be used at the exit interview after the last treatment, and a final time four weeks after the last treatment. This is because we are interested in the duration of potential benefit from acupuncture treatment.

Patients will be randomly assigned to one of two groups. All acupuncture will be performed through plastic shields so that the patient does not know which group he or she has been assigned to. In the first type of acupuncture, retractable needles are used such that the patient feels a pin sensation but there is no penetration of the epidermis. In the second type, non-retractable needles penetrate the acupuncture points into deeper tissue. It is not known whether deeper penetration is required for acupuncture to work, or if acupuncture is of benefit at all for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Symptomatic IC for at least six months
* Urinary frequency of at least eleven voids in a 24 hour period
* A self-rated global discomfort score of 4 or greater on a 0-10 scale

Exclusion Criteria:

Medical History or Co-Morbid Conditions:

* Any history of: bladder calculus, tuberculous cystitis; neurological disease or diabetic cystopathy; malignant bladder tumors, urethral cancer
* Prior 3 years of uterine, cervical or vaginal cancer (women only)
* Prior 6-12 weeks of: bacterial urinary tract infection; active genital herpes; gross hematuria
* Concurrent active urethral calculus, ureteral calculus, symptomatic urethral diverticulum; documented chronic bacterial prostatitis (men only); active vaginitis, pregnancy (women only)

Prior and Concurrent Treatment for IC:

* Any history of: cyclophosphamide, pelvic radiation; augmentation cystoplasty, cystectomy or cystolysis, neurectomy, implanted peripheral nerve stimulator; prostate surgery or treatment (men only)
* In the prior 24 weeks: any treatment with intravesical BCG, cystocele, rectocele, urinary incontinence surgery, transvaginal surgery, hysterectomy, prolapse, vaginal delivery or C-section (women only)
* Prior 6-12 weeks: any treatment by urethral dilatation, cystometrogram, urodynamics, cystoscopy/hydrodistention, bladder biopsy; prostate biopsy (men only); any intravesical treatment other than BCG
* Prior 4 weeks: any new medications initiated for IC
* Concurrent intravesical heparin, chronic use of acetylsalicylic acid, non-steroidal anti-inflammatory drugs or opioid pain medications for another pain condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Rate of improvement between arms as indicated by a Patient Overall Rating of Improvement Scale

SECONDARY OUTCOMES:
Improvement in Interstitial Cystitis Symptom and Problem Indices (validated symptom-specific measures)
Improvement in University of Wisconsin-Interstitial Cystitis Scale (validated symptom-specific measure)
Improvement in frequency, urgency and nocturia as measured on bladder diaries

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Pain Medicine Center, Philadelphia, Pennsylvania, United States